CLINICAL TRIAL: NCT01790477
Title: Auricular Acupuncture for The Treatment of Post-Tonsillectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2012.0102
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Recurrent Tonsillitis; Peritonsillar Abscess; Obstructive Sleep Apnea
Keywords: Tonsillectomy; Acupuncture
MeSH Terms: conditions — Tonsillitis; Peritonsillar Abscess; Sleep Apnea, Obstructive | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Auricular Acupuncture (Experimental): Use of auricular acupuncture in bilateral ears
  Interventions: Procedure: Auricular Acupuncture
- Control (No Intervention)

INTERVENTIONS:
Procedure: Auricular Acupuncture — Application of auricular acupuncture to 5 points on the ear
  Arms: Auricular Acupuncture

SUMMARY:
The goal of this study is to assess the role of battlefield acupuncture in the reduction of pain scores status post adult tonsillectomy. Secondary goals of this study include reduction in narcotic usage, decreased nausea and vomiting, and evaluating patient factors that lend an increased risk of worsening pain or improved response with acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who meets criteria and is scheduled for tonsillectomy

Exclusion Criteria:

* Any patient with prior use of acupuncture
* Individuals under age 18
* Tonsillectomy performed with other surgical procedures, i.e UPPP, adenoidectomy,
* Patients with a known personal or family history of a bleeding disorder will be excluded.
* Patients with a history of kidney or liver problems will also be excluded.
* Patients found to be pregnant will be excluded from participation.
* Patients unwilling to enroll in the study will have the tonsillectomy with or without adenoidectomy performed according to current practice standards.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Reduction in VAS scores between experimental and control group | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anil Shah, Principal Investigator — NMCSD
Locations (1):
- NMCSD Balboa, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No